CLINICAL TRIAL: NCT07225023
Title: A Multi-Site Feasibility Trial of Embedded Emergency Department Physical Therapy for Dizziness
Acronym: FEED-PT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: University of Utah (Other); Northwestern Lake Forest Hospital (Other); Northwestern Memorial Hospital (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Howard Kim, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FEED-PT for Dizziness; R21DC022877 (NIH)
Record Dates: First submitted 2025-10-10; First posted 2025-11-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Dizziness
Keywords: dizziness; Physical therapy; FEED-PT; Feasibility; Emergency Department
MeSH Terms: conditions — Dizziness; Emergencies

STUDY DESIGN:
Intervention Model Description: Two hospital EDs (Northwestern Memorial Hospital, University of Utah Hospital) will be randomized to receive either the embedded ED physical therapist intervention (treatment, n=1) or usual care (control, n=1). Following completion of the feasibility trial, the control site will receive the intervention as per standard waitlist procedures for randomized trials. A third hospital ED (Northwestern Lake Forest Hospital) will not participate in randomization or participant enrollment but will contribute electronic health record data to assist in feasibility assessments for a future full-scale trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Embedded Emergency Department Physical Therapy (Experimental): We place a physical therapist directly in the emergency department to initiate timely care for patients with dizziness rather than waiting on an outpatient referral to physical therapy, which can often take weeks to accomplish, if ever at all. The actual techniques and approaches used by the embedded ED physical therapist in this study (e.g., exercises, maneuvers, coaching) are standard-of-care and do not involve investigational interventions, devices, or drugs.
  Interventions: Other: Embedded Emergency Department Physical Therapy
- Usual Care (Other): Usual care treatment for dizziness presenting in the emergency department (ED). Usual care consists of any ED testing or treatment not involving an ED physical therapist in accordance with the treating physician's usual and customary practice. This could include diagnostic imaging, patient education and resources, and administration and/or prescribing of medications.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Embedded Emergency Department Physical Therapy — We place a physical therapist directly in the emergency department to initiate timely care for patients with dizziness rather than waiting on an outpatient referral to physical therapy, which can often take weeks to accomplish, if ever at all. The actual techniques and approaches used by the embedded ED physical therapist in this study (e.g., exercises, maneuvers, coaching) are standard-of-care and do not involve investigational interventions, devices, or drugs.
  Arms: Embedded Emergency Department Physical Therapy
Other: Usual Care — Standard-of-care treatment for dizziness presenting in the emergency department
  Arms: Usual Care

SUMMARY:
This is a multi-site feasibility trial of an embedded emergency department (ED) physical therapy care model for dizziness at two EDs in the Northwestern Medicine and University of Utah Health systems. The study intervention (embedded ED physical therapy) is a reconceptualization of the traditional outpatient physical therapy care model in which we place a physical therapist directly in the ED to initiate timely care for patients with dizziness; we previously evaluated this intervention in a single center randomized trial for low back pain. This multi-site feasibility trial will be comprised of 9 months of active intervention and 12 months of longitudinal data collection. The two sites will be parallel randomized 1:1 to receive either the embedded ED physical therapy condition (intervention, n=1) or usual care (control, n=1) via simple randomization. This trial focuses on feasibility outcomes - such as our ability to enroll participants, deliver the intervention with fidelity, and collect longitudinal patient-reported outcome data and electronic health record data.

DETAILED DESCRIPTION:
After a 12-month milestone-driven planning and preparation phase, we will conduct a 21-month randomized feasibility clinical trial of the embedded ED physical therapy intervention at the Northwestern Medicine and University of Utah health systems, comprised of 9 months of active intervention and 12 months of longitudinal data collection. Two hospital EDs (Northwestern Memorial Hospital, University of Utah Hospital) will be randomized to receive either the embedded ED physical therapist intervention (treatment, n=1) or usual care (control, n=1). Following completion of the feasibility trial, the control site will receive the intervention as per standard waitlist procedures for randomized trials. A third hospital ED (Northwestern Lake Forest Hospital) will not participate in randomization or participant enrollment but will contribute baseline electronic health record data to assist in feasibility assessments for a future full-scale trial.

ELIGIBILITY:
Inclusion Criteria:

* Emergency Department (ED) visit with primary diagnosis related to dizziness
* ED visit occurring at an ED site participating in randomization (Northwestern Memorial Hospital, University of Utah Hospital)
* ED visit check-in time during the hours of 8am-8pm
* Age greater than or equal to 18 years; there is no age maximum
* English or Spanish-speaking

Exclusion Criteria:

* Severe neurologic deficit concerning for ischemic or hemorrhagic stroke (i.e., that would necessitate activating a stroke code)
* Currently in police custody
* Unable to consent
* Known pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-09-06 (Estimated)

PRIMARY OUTCOMES:
Longitudinal participant surveys (effectiveness): missing data rate for the Dizziness Handicap Inventory | 12 months
  Rate of missing data for assessments administered between baseline and 12 months. Variable type: binary / proportion.
Longitudinal participant surveys (effectiveness): screening-to-enrollment ratio | Baseline
  Number of participants who enter screening compared to the number of participants who enroll in the study. Variable type: binary / proportion.
Longitudinal participant surveys (effectiveness): participant retention rate defined as completion of at least one follow-up survey. | 12 months
  Ratio of participants enrolled to the number who complete at least one follow-up survey.
Electronic Health Record (EHR) extraction (implementation): adoption of Emergency Department (ED) physical therapy | Baseline
  Adoption is defined as the number of potentially eligible dizziness ED visits have a documented order for a physical therapy evaluation. Cross-sectional at the level of site/Emergency Department during the trial. Variable type: Proportion.
Electronic Health Record (EHR) extraction (implementation): fidelity of Emergency Department (ED) physical therapy | Baseline
  Fidelity is defined as the number of dizziness ED visits that have a structured research note documenting use of the protocol. Cross-sectional at the level of site/Emergency Department (ED) during the trial. Variable type: proportion.
Clinician surveys before and after implementation of the intervention (implementation): Normalisation Measure Development Questionnaire (NoMAD) questionnaire scores | 1-6 months prior to opening study to accrual and 1-6 months after the last participant enrolls at the site.
  1-6 months prior to opening study to accrual and 1-6 months after the last participant enrolls at the site. Variable type: continuous.

SECONDARY OUTCOMES:
Longitudinal participant surveys (effectiveness): a sum of the missing data rate for the remaining Participant Reported Outcomes (PROs) combined. | 12 months
  Missing data rate for each PRO will not be analyzed separately, but will be combined into one measurement as one outcome. PROs: nine-item Vestibular Activities Avoidance Instrument (VAAI), Global Rating of Change, Numeric Pain Rating Scale, additional healthcare utilization (e.g., physical therapy, ED, doctor's office), and a medication use survey.
Electronic Health Record (EHR) extraction (effectiveness): rate of subsequent health care encounters. | 12 months
  Variable type: count, may be considered binary / proportion
Electronic Health Record (EHR) extraction (effectiveness): rate of prescribing sedating medications (including antihistamines and benzodiazepines) | 12 months
  Variable type: count, may be considered binary / proportion
Electronic Health Record (EHR) extraction (effectiveness): rate of advanced diagnostic imaging | 12 months
  Variable type: count, may be considered binary / proportion
Clinician surveys before and after implementation of the intervention (implementation): Acceptability of Intervention Measure (AIM) | 1-6 months prior to opening study to accrual and 1-6 months after the last participant enrolls at the site.
  1-6 months prior to opening study to accrual and 1-6 months after the last participant enrolls at the site. Variable type: continuous. Minimum value is 4, Maximum value is 20. Higher scores = higher agreement with outcome.
Clinician surveys before and after implementation of the intervention (implementation): Intervention Appropriateness Measure (IAM) | 1-6 months prior to opening study to accrual and 1-6 months after the last participant enrolls at the site.
  1-6 months prior to opening study to accrual and 1-6 months after the last participant enrolls at the site. Variable type: continuous. Minimum value is 4, Maximum value is 20. Higher scores = higher agreement with outcome.
Clinician surveys before and after implementation of the intervention (implementation): Feasibility of Intervention measure (FIM). | 1-6 months prior to opening study to accrual and 1-6 months after the last participant enrolls at the site.
  1-6 months prior to opening study to accrual and 1-6 months after the last participant enrolls at the site. Variable type: continuous. Minimum value is 4, Maximum value is 20. Higher scores = higher agreement with outcome.

OTHER OUTCOMES:
Participant and clinician focus groups (implementation) | 1-6 months before the first participant enrolls and 1-6 months after the study closes to follow-up.
  These data will be collected and analyzed qualitatively.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Scientific data and metadata will be archived into Northwestern University Libraries' institutional repository, Arch (https://arch.library.northwestern.edu/). Northwestern University faculty, students, and staff with a current NetID are allowed unlimited storage, file uploads, and hosting for their scientific work.
  Scientific data will be made available at the end of the award period or at the time of the corresponding publication, in the case of any publications that pre-date the award end date. Datasets resulting from this work will remain available in the repository in perpetuity or until deaccessioned at the discretion of the repository. Should the funding or organizational imperatives of the Northwestern University Libraries change, the Libraries will strive to provide at least one year notice, and devote resources to support the transition to another host institution and/or returning the data to the data producers.
Supporting Information: Study Protocol, SAP
Time Frame: Scientific data will be made available at the end of the award period or at the time of the corresponding publication, in the case of any publications that pre-date the award end date. Datasets resulting from this work will remain available in the repository in perpetuity or until deaccessioned at the discretion of the repository.
Access Criteria: Access to scientific data and metadata will not be controlled after archiving. Arch is an open access repository that is focused on digital data archiving and unmediated public access to research results.